CLINICAL TRIAL: NCT05396768
Title: Validation of a New Assessment Tool for Chest Tube Insertion (ACTION) on Two Different Simulators
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10905
Record Dates: First submitted 2022-05-16; First posted 2022-05-31 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Educational Assessment; Chest Tube Insertion; Validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novices: Junior residents from the departments of surgery, pneumology or emergency medicine. These participants are in their first or second year of residency, and have observed or placed less than 5 CTIs in their career.
  Interventions: Other: Assessment using the ACTION-tool.
- Experienced: Faculty members from Ghent University Hospital from the departments of surgery, pneumology or emergency medicine. These participants must have finished their residency training, and must be involved in resident education.
  Interventions: Other: Assessment using the ACTION-tool.

INTERVENTIONS:
Other: Assessment using the ACTION-tool. — Participants will be assessed using the ACTION-tool while they are performing a CTI on a porcine rib model and Thiel embalmed human cadavers.

SUMMARY:
The aim of this study is to collect validity evidence for the ACTION-tool on two different simulators: a porcine rib model, and Thiel embalmed human cadavers. Validity evidence will be collected following Messick's framework.

DETAILED DESCRIPTION:
Educational assessments need a validity argument before they are being used to evaluate trainees. An assessment needs to show it can be used as an objective and reliable tool.

Messick's framework of validity collects this evidence from five different sources: content, response process, relation to other variables, internal structure and consequences.

The ACTION-tool has been developed based on a Delphi consensus study (and has established content evidence as a result). This study will collect evidence from the four remaining sources.

Two groups of participants (novices and experienced) will be recruited. All participants will provide informed consent and demographic information. Afterwards, they will be informed of the study, will familiarise themselves with the simulators, watch an educational video, and will be asked to perform two chest tube insertions (CTI).

All participants will be evaluated by a live rater, and will be recorded using a head-mounted GoPro and an overview camera. The recordings will be edited to ensure anonymization, and will be subsequently rated by three blinded raters.

Statistical analysis will evaluate the difference in mean scores between the groups, the internal structure using G-theory, and will establish a pass/fail score.

ELIGIBILITY:
Inclusion Criteria:

* Experienced participants must hold a degree of Master in Medicine, and must have finished the residency training specific to their field (attending physician).
* Novice participants are defined as junior residents who are graduated as Master in Medicine and must be in their first two years of residency training, or be at least in their 3rd Master year of Medicine and be accepted as starting resident.

Exclusion Criteria:

* Experienced participants who lack experience or the appropriate diplomas will be excluded.
* Novices who have performed more than five CTI or assisted in the placement of more than five procedures will be excluded.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from Ghent University Hospital. Experienced participants are faculty members, and the novice group is recruited from the resident population.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Score on on the ACTION-tool | Immediately after performing a CTI on the simulator.
  The main goal is the collection of validity evidence for the ACTION-tool following Messick's framework. This is done by recording the score each participant receives while being assessed using the ACTION-tool. The minimum score on the rating scale is 17, the maximum 85 (a higher score indicates a better performance). On the error checklist the minimum score is 0, maximum score is 16 (where a lower score is less observed errors).

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Willaert, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No